CLINICAL TRIAL: NCT05041491
Title: Breaking up Sedentary Time to Improve Glucose Control in a Population at Risk for Developing Type 2 Diabetes
Acronym: BURST2D
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-1900
Record Dates: First submitted 2021-08-26; First posted 2021-09-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pre-diabetes
Keywords: sedentary behavior; physical activity; glucose control; metabolism; pre-diabetes
MeSH Terms: conditions — Glucose Intolerance; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the BREAK condition (5-min bouts of brisk walking performed hourly for 9 hours/day, 5 days/wk) or the ONE condition (45-min of brisk walking performed as a single continuous bout, 5 days/wk) for 3 months. Participants will complete all study visits in only one group.
Who Masked: Outcomes Assessor
Masking Description: A study research assistant that is not involved in the study participants' allocation process will create opaque, sealed envelopes with allocation sequences based on the randomization table created by the study statistician. The assignment of intervention to study participants will be based on the study allocation sequence generated by the statistician and the study team will enroll study participants and assign them to the interventions. The study team will be blinded until study participants' allocation (the day before visit G). After this, the study team will not be blinded to study participants' allocation as they will be responsible for assigning study participants, and for applying and monitoring the interventions. The study statistician will always be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREAK Intervention (Experimental): Participants in the BREAK condition will perform 5-minute bouts of brisk walking hourly for 9 hours/day, 5 days/week for 3 months.
  Interventions: Behavioral: BREAK
- ONE Intervention (Active Comparator): Participants in the ONE condition will perform 45 minutes of brisk walking as a single continuous bout, 5 days/week for 3 months.
  Interventions: Behavioral: ONE

INTERVENTIONS:
Behavioral: BREAK — The BREAK intervention is a physical activity regimen.
  Arms: BREAK Intervention
Behavioral: ONE — The ONE intervention is a physical activity regimen.
  Arms: ONE Intervention

SUMMARY:
Newly released guidelines recommend increased physical activity (PA) and reduced sedentary behaviors (SB) to improve glycemia and prevent the onset and progression of type 2 diabetes (T2D). Typically, 30-60 min bouts of PA are advocated per day. Although this approach increases PA, it does not decrease the length of the sedentary periods through the day. This is important because recent epidemiological data suggest that frequently interrupting sedentary time improves glucose control even in people who achieve the recommended levels of PA. Preliminary experimental data suggest that breaking up prolonged sedentary time by performing multiple short bouts (5 min) of PA throughout the day, may improve glycemia more than performing a single continuous bout of PA, and thereby potentially be a novel strategy to prevent T2D. The improvement in glycemia was observed even when the total amount of PA and total energy expenditure were matched, suggesting that how and when PA is performed over the day may matter more than how much PA is done. However, important gaps in knowledge remain including: (1) whether similar benefits on glucose control would be observed in adults with prediabetes, a clinically relevant population that is at high risk of developing T2D; (2) whether these effects are sustained or diluted over time, and (3) what are the mechanistic underpinnings. To address these gaps, the investigators propose to measure the acute and chronic effects of PA breaks on glucose control and the underlying mechanisms in individuals at risk of developing T2D. Sedentary men and women with prediabetes (n=66, 50% F) will be randomized to either an intervention designed to interrupt SB with 5-min bouts of brisk walking performed hourly for 9 hours/day, 5 days/week (BREAK) or a control condition consisting of 45-min of brisk walking performed as a single daily continuous bout, 5 days/week (ONE). The two 3-months interventions will be matched for total active time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* BMI of 18.5-40 kg/m2 and weight stable over the previous 6 months.
* Age, 18-64 years old.
* Fasting glucose of 100-125 mg/dL or fasting HbA1c of 5.7-6.4%, or 2h OGTT blood glucose of 140-199mg/dL based on the American Diabetes Association criteria for pre-diabetes. Fasting glucose, HbA1c and OGTT results ordered by the participant's provider within 3-months of the screening visit will be accepted, provided they fall within the measurement of error range established by the institution's lab standards. Additionally, consistent use of Metformin (1 year) to prevent prediabetes from developing diabetes will be accepted.
* Less than 150 minutes of moderate-to-vigorous physical activity (MVPA) per week and more than 6 hours of sitting time per day, as self-reported by the volunteers using the International Physical Activity Questionnaire (IPAQ).
* Less than 6500 of steps per day as measured by a pedometer over 5 days (at least 1 weekend day).
* Passing medical and physical screening, and analysis of blood and urine screening samples.
* Low-moderate caffeine use (<3 cups/day).
* Agree to refrain from any other structured exercise than the physical activity prescribed in each arm of the study.
* Agree to eat control diets for 3 days before and during the Clinical and Translational Research Center (CTRC) visits;
* Agree to refrain from taking any over-the-counter (including nonsteroidal anti-inflammatory drugs) or prescribed medication (apart from oral contraceptives) for 3 days prior to the inpatient CTRC visits;
* Agree to wear a Fitbit® activity monitor and upload data on the website on a daily basis for the whole duration of the study.
* Agree to follow the physical activity interventions and to be randomly assigned to one of the two arms of the study.
* Agree to complete all the study procedures.

Exclusion Criteria:

* Pregnancy, breast-feeding or post-menopause for women.
* Being considered unsafe to participate as determined by the study physician.
* Ever having a history of systemic, psychiatric, neurological disease, or drug and alcohol abuse.
* History of cardiovascular disease, diabetes, uncontrolled hypertension, untreated thyroid, renal, hepatic diseases, dyslipidemia or any other medical condition affecting weight or lipid metabolism.
* Being positive for human immunodeficiency virus or hepatitis B or C.
* Taking medications affecting weight, triglycerides, energy intake/energy expenditure, or sleep in the last 3 months.
* Having abnormal blood chemistry and/or hematology as deemed significant by the study physician.
* Being a smoker or having been a smoker in the 3 months prior to their screening visit.
* Having donated over 400 mL of blood within 3 months (90 days) of screening for the study;
* Working night shifts within 1 month of and throughout the study.
* Not completing the trial days of BREAK and ONE during the screening period to assess the willingness and ability of the participant to perform each of the interventions.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Glycemia | Glucose concentration in mg/dl, measured at fasting, during a 2 hour OGTT and after
  Plasma glucose concentration in mg/dL measured before and 30, 60, 90 and 120 min after an oral glucose tolerance test (OGTT, 75g glucose).

SECONDARY OUTCOMES:
Insulinemia | Plasma insulin concentration in mUI/mL, measured at fasting, during a 2 hour OGTT and after
  Plasma insulin concentration in milli-international units per milliliter (mUI/mL) measured before and 30, 60, 90 and 120 min after an oral glucose tolerance test (OGTT, 75g glucose).
Mean interstitial glucose concentration | Before and after 1 month and 3 months of intervention
  Mean interstitial glucose concentration measured continuously by a glucose monitor placed on the tricep for 24hours for 10 days.
Daily glycemia variability | Before and after 1 month and 3 months of intervention
  Standard deviation (SD) of interstitial glucose concentration measured continuously by a glucose monitor placed on the tricep 24hours throughout 10 days.
Fasting A1c concentration | Time Frame: Before and after 1 month and 3 months of intervention
  Fasting A1c concentration expressed in %
Fasting fructosamine concentration | Before and after 1 month and 3 months of intervention
  Fasting fructosamine concentration in umol/L
12-hour exogenous glucose oxidation | Before and after 1 month of intervention
  Rates of carbon-13 (13C) recovery (% of the dose) in expired carbon dioxide (CO2) following the ingestion of U-13C-glucose in both breakfast and lunch meals.
12-hour endogenous glucose oxidation | Before and after 1 month of intervention
  Rates of D2 recovery (% of the dose) in expired urines following the infusion of (2,2H2) glucose.
12 hour CO2 production | Before and after 1 month of intervention
  CO2 production measured by indirect calorimetry (ParvoMedics TrueOne® 2400, Salt Lake City) for 20 minutes every hour from 0800h to 1800h.
12 hour O2 production | Before and after 1 month of intervention
  O2 production measured by indirect calorimetry (ParvoMedics TrueOne 2400, Salt Lake City) for 20 minutes every hour from 0800h to 1800h.
12 Urine excretion | Before and after 1 month of intervention
  Urine will be measured every hour from 0730h to 1830h
Glucose kinetics | Before and after 1 month of intervention
  Steele's equation for non-steady-state will be used to compute rate of appearance of total glucose (RaT) and rate of appearance of exogenous glucose (RaE), as well as the rates of disappearance (RdT and RdE) from the percentage of [6,6-2H2]glucose6 and of 13C-glucose in plasma glucose61. Endogenous glucose production (EGP) will be computed as RaT-RaE. Nonoxidative glucose disposal (NOGD) will be calculated by subtracting total carbohydrate oxidation from (RdT + RdE). Plasma glucose utilization will be assumed to be equivalent to RdT as has been confirmed previously. Muscle glycogen utilization during the active period will be calculated as total carbohydrate utilization during exercise minus plasma glucose utilization during exercise.
Fasting and postprandial glucose | Before and after 1 month of intervention
  Fasting and postprandial glucose in mg/dl measured in response to standard lunch
Fasting and postprandial insulin | Before and after 1 month of intervention
  Fasting and postprandial insulin in ml/iu measured in response to standard lunch
Fasting and postprandial C-Peptide | Before and after 1 month of intervention
  Fasting and postprandial C-peptide nmol/mL measured in response to standard lunch
Fasting and postprandial glucagon | Before and after 1 month of intervention
  Fasting and postprandial glucagon in pg/mL measured in response to standard lunch
Fasting and postprandial catecholamines | Before and after 1 month of intervention
  Fasting and postprandial catecholamines in pg/mL measured in response to standard lunch
Skeletal muscle content of protein kinase B (Akt) (Aktser473/total) | Before and after 1 month of intervention
  Vastus lateralis skeletal muscle biopsies will be collected from fasting participants by the Bergstrom technique. Biopsies will be used to measure protein kinase B (Akt) (Aktser473/total) using western blotting.
Skeletal muscle content of ACC (ACCS79/ total) | Before and after 1 month of intervention
  Vastus lateralis skeletal muscle biopsies will be collected from fasting participants by the Bergstrom technique. Biopsies will be used to measure ACC (ACCS79/ total) using western blotting.
Skeletal muscle content of TBC1D4 (AS160/ total) | Before and after 1 month of intervention
  Vastus lateralis skeletal muscle biopsies will be collected from fasting participants by the Bergstrom technique. Biopsies will be used to measure TBC1D4 (AS160/ total) using western blotting.
Skeletal muscle content of COX4 | Before and after 1 month of intervention
  Vastus lateralis skeletal muscle biopsies will be collected from fasting participants by the Bergstrom technique. Biopsies will be used to measure citrate synthase (COX4) using western blotting.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Bergouignan, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No